CLINICAL TRIAL: NCT00438035
Title: Evaluation of Postoperative Pain by Spectral Analysis of ECG R-R Intervals
Brief Title: Heart Rate Variability and Postoperative Pain
Acronym: ECG-Spectral
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2002
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2007-02

CONDITIONS: Pain; Postoperative
Keywords: Postoperative pain; Heart rate variability, sympathetic, parasympathetic; Visual analog pain scale; Spectral analysis of ECG
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ECG spectral

SUMMARY:
Postoperative pain stimulates the autonomic nervous system, induces the production of pro-inflammatory substances, reduces patient mobility and impairs vital functions. The ECG spectral analysis (ECGs) is a non-invasive marker of the autonomic nervous system state. To our knowledge, the correlation between the sympathovagal activity quantified by a non invasive method and the postoperative pain, has not been studied before.

DETAILED DESCRIPTION:
* Principal Objective : 1)To quantify postoperative pain by the ECGs technique. 2) To compare the ECGs parameters with the visual analog pain scale (VAS) results.
* Secondary Objective : To determine the influence of preoperative chronic pain and pathophysiological profiles on the correlation between postoperative ECGs and VAS.
* Study design : An observational, prospective, single arm, single center study.
* Inclusion criteria : ¨Patients over 18 years old scheduled for surgery under general anesthesia. Patients capable of using the visual analog pain scale.
* Exclusion criteria : Pregnancy or breast feeding, impossibility to obtain an informed consent, incapacity to follow all the study schedule. Patient not protected by social security, patient likely to present hypovolemia or severe hemodynamic instability. Patient with a dysautonomia characterized by orthostatic hypotension, patients with cardiac disarrhythmias, likely to interfere with the ECG and/or the spectral analysis of ECG.
* Study plan: Patients will sign their informed consent during the V0 visit (preoperative). During V0, HF and LF (ECGs parameters) will be measured as well as the VAS-estimated pain. These results, medical history, concomitant diseases and medications will be reported in a case report form (CRF). The second and last visit, V1, takes place 1 hour after the patient wakes up, in the postoperative period. ECGs and VAS evaluation will be achieved in the same manner as the V0 visit. The only difference is that the measurements will be repeated to obtain a total of 5 data couples over 2 hours. These Intrapatient estimations will be used to improve statistical ECGs vs VAS correlation analysis.
* Number of subjects : 100

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old scheduled for surgery under general anesthesia.
* Patient able to use the visual analog pain scale

Exclusion Criteria:

* Pregnancy or breast feeding
* Impossibility to obtain an informed consent
* Incapacity to follow all the study schedule
* Patient not protected by social security
* Patient likely to present hypovolemia or severe hemodynamic instability
* Patient with a dysautonomia characterized by orthostatic hypotension
* Patient with cardiac disarrhythmias, likely to interfere with the ECG and/or the spectral analysis of ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Spectral ECG | Preoperative and postoperative time

CONTACTS AND LOCATIONS:
Overall Officials: Musa SESAY, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Neurochirurgie A, hôpital Pellegrin, Bordeaux, Place Amélie Raba-Léon, France

REFERENCES:
- [Background] Sesay M, Vignes JR, Liguoro D, Crozat P, Boulard G, Guerin J, Barat M, Maurette P. [Autonomic hyperreflexia induced by sacral root stimulation is detected by spectral analysis of the EEG]. Can J Anaesth. 2002 Nov;49(9):936-41. doi: 10.1007/BF03016878. French. PMID 12419720
- [Derived] Sesay M, Robin G, Tauzin-Fin P, Sacko O, Gimbert E, Vignes JR, Liguoro D, Nouette-Gaulain K. Responses of heart rate variability to acute pain after minor spinal surgery: optimal thresholds and correlation with the numeric rating scale. J Neurosurg Anesthesiol. 2015 Apr;27(2):148-54. doi: 10.1097/ANA.0000000000000102. PMID 25105826